CLINICAL TRIAL: NCT03262532
Title: Assessment of a Web-Based Simulation Module to Improve Performance in Obtaining Standard Transesophageal Echocardiography (TEE) Views
Brief Title: Assessment of a Web-Based Simulation in Transesophageal Echocardiography (TEE) Views
Acronym: Web-SimTEE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: REB 15-9547
Record Dates: First submitted 2017-03-30; First posted 2017-08-25 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2017-11

CONDITIONS: Education; Training
Keywords: Interactive web-base simulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: Learning TEE manipulation with a Web-based TEE simulation module
  Interventions: Other: Web-base simulator
- Control: Learning a TEE manipulation without the Web-based TEE simulation
  Interventions: Other: No web-base simulator

INTERVENTIONS:
Other: Web-base simulator — Training manipulation of TEE using a Web-based simulator
  Groups: Experimental
Other: No web-base simulator — Training manipulation of TEE with out a web-base simulator
  Groups: Control

SUMMARY:
Transesophageal echocardiography (TEE) is often used by anesthesiologists during cardiac surgery, as a monitoring tool in non-cardiac surgery, and as a point of care diagnostic tool in the intensive care unit (ICU). Furthermore, TEE is becoming a core skill in many specialties to facilitate focused cardiovascular assessment in hemodynamically compromised patients in various settings. Educators must determine how to best instruct current and future trainees to achieve clinical competence in TEE within a time limited and constantly expanding medical curriculum.

In this study the investigators will evaluate a new online TEE Simulation module as a learning tool to accelerate and enhance traditional clinical teaching. This project will evaluate a new online TEE Simulation module that replicates the actions required to adjust TEE probe position and the ultrasound plane in relation to a 3D heart model.

The investigators hypothesize that experience with the online TEE simulation module will improve the ability of trainees to independently perform TEE probe manipulations necessary to obtain standard TEE views. The proposed study will answer this question by measuring the performance of trainees in obtaining 10 of the 25 standard TEE views using the Vimedix mannequin-based ultrasonography simulator following an hour of review of the online TEE Simulation module.

The educational benefit of the Web-based TEE simulation module, will be evaluated by 20 novices randomly assigned to two groups, a control group of 10 subjects without exposure to the Web-based simulation, and an experimental group of 10 subjects with exposure to the Web-based simulation. Both groups will be assessed on their performance in attaining the 10 standard TEE views with the Vimedix simulator.

ELIGIBILITY:
Inclusion Criteria:

* Residents or fellows in anesthesia, cardiology and critical care enrolled at the Toronto General Hospital

Exclusion Criteria:

* Residents or fellows in anesthesia, cardiology and critical care with prior experience with TEE probe manipulation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will recruit residents and fellows during their training from the University of Toronto postgraduate programs in anesthesia, cardiology and critical care. They will have some knowledge of transthoracic echocardiography but no prior experience with TEE probe manipulation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-07-01 (Estimated); Study Completion 2018-09-01 (Estimated)

PRIMARY OUTCOMES:
TEE simulation model decreases time to select image acquisition in trainee participant vs. participants trained by reading material only | 2 week review 1 session for assessment (Control: time required to acquire 10 views, Intervention: I hour session with online simulator plus time required to acquire 10 views)
  The metrics for acquiring each image will be recorded by the model, the primary measurement will be time in seconds per view acquired.

SECONDARY OUTCOMES:
TEE simulation model improves select image quality in trainee participants vs. participants trained by reading material only as assessed by a expert review panel of echo cardiographers | 2 week review 1 session for assessment- time required to acquire 10 views
  Each image will be captured by the model and graded according to a 5 point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Publication